CLINICAL TRIAL: NCT00475748
Title: ASIA Motor, Functional and Health Related Quality of Life Outcome in Traumatic Central Cord Syndrome, a Prospective Randomized Study
Brief Title: Surgical Management of Spinal Cord Injuries In Neck
Acronym: CCSS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Maryland Department of Health and Mental Hygiene (Other Government)
Collaborators: University of Maryland, Baltimore (Other)
Responsible Party: Bizhan Aarabi, University of Maryland
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-28962; Maryland DHMH# FHA07-004
Record Dates: First submitted 2007-05-17; First posted 2007-05-21 (Estimated); Last update posted 2009-06-24 (Estimated); Status verified 2009-06

CONDITIONS: Central Cord Syndrome; Spinal Cord Injury; Quadriparesis
Keywords: cervical spine; spinal cord; trauma; spinal cord injury; central cord syndrome
MeSH Terms: conditions — Central Cord Syndrome; Spinal Cord Injuries; Quadriplegia; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Early and late surgery for traumatic central cord syndrome — Surgical decompression of the spinal cord, either front, back or combined

SUMMARY:
ABSTRACT/EXECUTIVE SUMMARY BACKGROUND, SIGNIFICANCE & RATIONALE: Between 10-20% of the more than 6000 cases of spinal cord injury seen annually in the North America have the clinical pattern of traumatic central cord syndrome (TCCS). These patients are usually older, most likely have sustained a fall, and have incomplete spinal cord injury characterized by dysesthetic and weak upper extremities. CT scan of the cervical spine in patients with TCCS often shows disc/osteophytes complex superimposed on degenerative or congenital spinal stenosis and MRI reveals signal changes at one or multiple skeletal segments. A minority of these patients suffer from fracture/subluxations, however, this group of patients are younger and have been involved in a more dynamic trauma. Since 1951, when Schneider et al reported this syndrome, controversy has dominated its surgical management. The current "Guidelines for the Management of Acute Cervical Spine and Spinal Cord Injuries" recommendations are only at the level of options, since prospective outcome data are unavailable.

HYPOTHESIS: in acute traumatic central cord syndrome, surgical decompression of the spinal cord within five days will result in more rapid motor recovery, than decompression 6 weeks following injury. To test this hypothesis, we will pursue the following specific aims:

SPECIFIC AIM I: To compare American Spinal Injury Association (ASIA) Motor Scores after three months post injury in patients with central cord syndrome operated on within five days of injury to a similar group of patients operated on 6 weeks following injury.

SPECIFIC AIM II: To compare functional outcome, health related quality of life and posttraumatic syrinx size in patients with traumatic central cord syndrome operated on within five days to a similar group of patients operated on 6 weeks following injury.

DESIGN: Single center prospective randomized study. PROCEDURE: In a two-year period thirty patients with traumatic central cord syndrome and cord compression (15 patients in each group) will be randomized to undergo surgical decompression either within the first five days or at 6 weeks following spinal cord injury. ASIA motor, functional recovery and health related quality of life between the two groups will be compared at admission, discharge from rehab facility 3 months and 12 months after surgery.

DETAILED DESCRIPTION:
JUSTIFICATION Between 10-20% of the more than 6000 cases of cervical spinal cord injury seen annually in the North America have the clinical pattern of traumatic central cord syndrome (TCCS) . These patients are usually older, most likely have sustained a fall, and have incomplete spinal cord injury characterized by dysesthetic and weak upper extremities. CT scan of the cervical spine in patients with TCCS often shows disc/osteophytes complex superimposed on degenerative or congenital spinal stenosis and MRI reveals signal changes at one or multiple skeletal segments. A minority of these patients suffer from fracture/subluxations, however, these patients are younger and have been involved in a more dynamic trauma. Since 1951, when Schneider et al reported this syndrome, controversy and confusion has dominated its surgical management. The current "Guidelines for the Management of Acute Cervical Spine and Spinal Cord Injuries" recommendations are only at the level of options, since prospective outcome data are unavailable .

During the past four decades, there has been significant progress in our understanding of the pathophysiological mechanisms governing traumatic spinal cord injury including central cord syndrome. Translation of kinetic energy, primarily through hyperextension and less often fracture dislocations of cervical spine, usually involved with cervical spondylosis or congenital spinal stenosis, results in anatomical compression of the spinal cord followed by secondary insults which are time dependent and likely ischemic in nature. Microangiographic studies of spinal cord in patients with cervical spondylosis have indicated deformation, stretching and flattening of the spinal cord tracts as well as sulcal microvasculature, which may be further jeopardized by traumatic hyperextension, resulting in axonal interruption, swelling and vascular damage, predisposing to sustained spinal cord ischemia responsible for clinical manifestations of central cord syndrome.

HYPOTHESIS: in acute traumatic central cord syndrome, surgical decompression of the spinal cord within 1-5 days will result in more rapid motor and functional recovery and results in a better quality of life than decompression ~6 weeks following injury. To test this hypothesis, we will pursue the following specific aims: SPECIFIC AIM I: To compare American Spinal Injury Association (ASIA) Motor Scores after three and 12 months post injury in patients with central cord syndrome operated on within 1-5 days of injury to a similar group of patients operated on ~6 weeks (range 5-7 weeks) following trauma. SPECIFIC AIM II: To compare functional outcome, health related quality of life and posttraumatic syrinx size three and 12 months after injury in patients with traumatic central cord syndrome operated on within 1-5 days to a similar group of patients operated on ~6 weeks (5-7 weeks) following injury.

DESIGN/PROCEDURE Our investigation will be single center prospective randomized pilot study. Thirty conscious adult (>17 years old) patients with clinically (conventional ASIA exam) and radiologically (conventional MRI and CT of neck) proven cervical traumatic central cord syndrome will be screened for this study. These patients are admitted to the University of Maryland Medical System within 48 hours of their injury and are randomized (computer) into two surgical groups. Study subjects are fully resuscitated, stable and eligible to sign consent to go through the research process. None of these patients have radiologically overt unstable cervical spine injuries or any injury requiring urgent surgical decompression and stabilization. A computer designed random number generator will divide these patients into two standard of care surgical groups: Early Surgical Decompression Group ((ESDG [odd #])) will have surgery 1-5 days after trauma and the late surgical decompression group ((LSDG [even #])) will be operated after a period of ~ 6 weeks (range 5-7 weeks). Unless medically indicated to stay in an acute care facility, the LSD Group patients are discharged to a rehab facility or home to be brought back for surgery. While in hard collar the latter group will be studied with a CT of the neck at 3 weeks (designed as a research tool) in order to assure no missed ligamentous injury resulting in glacial instability. If hidden instability is discovered, depending on its severity, decompression and internal fixation may be performed earlier than the proposed 6 weeks. Both groups will have detailed conventional medical, neurological and radiological examination during their hospital stay and while in a rehab center, at 3 months, 6 months and 12 months postinjury. All the studies will be clinically conventional except MRI at 12 months post injury which is research related to measure the size of spinal cord syrinx. While ready to be discharged from a rehab center and at 3 and 12 months post injury all these patients will have detailed research related functional studies as depicted in study schedule in form of known outcome measures (Functional Independence Measure, Spinal Cord Independence Measure, and Walking Index for Spinal Cord Injury). In this study there won't be a placebo or control group.

Procedure

1. PREHOSPITAL ,Trauma Resuscitation Unit (TRU) & Emergency Department (ED) RESUSCITATION: In a two-year period, all patients admitted to the STC TRU and UMMS EDs, within 48 hours of their spinal cord injury, will be screened for evidence of acute traumatic central cord syndrome (TCCS).
2. SCREENING: Patients with incomplete spinal cord injury and MRI evidence of spinal cord compression and swelling are visited for a complete conventional American Spinal Injury Association Neurological and Functional Classification of motor, and sensory deficits. Those with ASIA Impairment Grades B, C and D/E and with the clinical picture of central cord syndrome will be chosen for possible enrollment. Inclusion/Exclusion Check List is by now complete.
3. RANDOMIZATION: We (PI or his designee) will use one of the computer programs to generate random numbers in order to divide 30 patients into two groups of surgical candidates (Nregnow/digital river Chicago IL 60695-0001). Odd numbers are used for early (1-5 days) decompression and even numbers for late ((after 6 weeks[5-7 weeks])) decompression. The software is set in such a manner so that only a single number is generated for a single patient with a specific alphanumerical user code (CCSS3001-CCSS3030). Generation of a random number is accomplished by the PI or his designee. Randomization is part of research process.
4. TIMING OF DECOMPRESSION: Based on the feasibility studies of Tator et al in STASCIS 1(please see the res of protocol), we decided to set the timing of decompression at five days (1-5 days) and six weeks (5-7weeks) in order to be able to capture most of the eligible patients. Enrollment will be within 48 hours of the injury. If due to any reason(s) (e.g. complications) a patient who is randomized for early surgery does not get operated, still he is followed as "an intent to treat patient" and his/her outcome will be analyzed. The same is true for a patient who is to have late surgery but due to a specific reason his surgery is cancelled.
5. OPERATIVE INTERVENTION: Eligible patients with traumatic central cord syndrome, canal compromise and spinal cord compression will be consented, and randomized into two groups. Thirty patients (15 patients in each group) will undergo standard surgical decompression of spinal cord either within the first five days or at 6 weeks following spinal cord injury. Each of the 15 patients enrolled for late decompression will be kept in hard collar while in a rehab facility and will undergo research related CT studies at 3 weeks post admission. If interim imaging studies indicate glacial translation, earlier decompression and internal fixation may be considered. The choice of surgical technique for decompression is standard of treatment at the Shock Trauma Center. Standard surgical decompression of the spinal cord will be by a select group of Department of Neurosurgery staff with full familiarity with cervical spine surgical interventions.
6. FOLLOW-UP OF PATIENTS: Before, immediately after and at 72 hours following surgery, at discharge from acute care or rehab center, 6 weeks, 3, 6, and12 months post injury patients will have complete conventional ASIA motor and sensory classification examination. Patients enrolled in the early surgical group will stay in the critical care or intermediate care unit, or the general floor until discharge to a rehabilitation center. These patients will have conventional postoperative CT while inpatient, at 3 and 12 months post injury. A research related CT (at 3 weeks) is performed in late surgery group in order to evaluate the stability of the sagittal plane of the cervical spine. Conventional MRI is performed before and immediately following surgery in every patient of the study and at 12 months (research related MRI) to evaluate the size of the spinal cord syrinx. SF-36, Functional Independence Scale (FIM), Walking Index for SCI (WISCI), Spinal Cord Independence Measure (SCIM), will be checked as an outcome measure research instrument at discharge from rehab facility, at 3 months, and at 12 months following injury in all patients. Patients randomized to have decompression at 6 weeks will have external fixation with a hard collar and will be transferred to a rehabilitation center or home for six weeks and then brought back for surgical decompression. Follow-up of these patients will be identical to the early operative group.
7. OUTCOME INSTRUMENTS American Spinal Injury Association Motor Score Classification: ASIA Motor Score. American Spinal Injury Sensory Score Classification: ASIA Sensory Score. ASIA impairment Score (A, B, C, D, E) Functional Independence Measure (FIM) Spinal Cord Independence Measure (SCIM). Walking Index of Spinal Cord Injury (WISCI). Health Related Quality of Life measure SF-36. CT evaluation of cervical spinal cord injury according to Allen-Ferguson Mechanistic Classification. CT quantification of canal compromise according to the formula of Fehlings et al. MRI evidence of spinal cord compression damage and syrinx size at specified intervals.

ELIGIBILITY:
Inclusion Criteria:

1. All adult patients (>17 years old) admitted to University of Maryland Medical System with traumatic central cord syndrome and evidence of spinal cord compression.
2. Allen-Ferguson Injuries: Distractive Extension Stages 1, Compressive Extension Stage 1, Vertical Compression Stages 1, Compressive Flexion Stage 1.
3. Patient with ASIA (American Spinal Injury Association) level of injury from C4 to T1 inclusive
4. Patients with ASIA (American Spinal Injury Association) Impairment Grades B, C, and D/E
5. Pregnant women 6-Lactating women

Exclusion Criteria:

1. Children aged <18
2. Terminally ill patients, patients with non-survivable injuries and patients with demyelinating disease.
3. Patients likely not to be able to appear for follow up.
4. Allen-Ferguson Injuries: Distractive Extension Stage 2, 3, Distractive Flexion Stages 1-4, Compressive Extension Stages 2-4, Vertical Compression Stages 2-4, Compressive Flexion Stages 2-4, Vertical Distraction Injuries.
5. Patients with acute disc herniation in need of urgent decompression.
6. Patients with progressive neurologic worsening
7. Patients with spinal cord injury without radiological abnormality (SCIWORA)
8. Central cord syndrome in association with traumatic brain injury (GCS<15)
9. Patients with previous cervical spine injury and /or surgery. 10-ASIA (American Spinal Injury Association) grade A patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-05; Primary Completion 2009-05 (Actual); Study Completion 2010-05 (Estimated)

PRIMARY OUTCOMES:
To compare ASIA Motor score after 3 months in patients with central cord syndrome operated on within five days to a similar group of patients operated on 6 weeks following injury. | one year
ASIA Motor Score | 12 months

SECONDARY OUTCOMES:
To compare functional outcome and quality of life at 3 and 12 months after injury 2) To compare the degree of canal compromise, spinal cord compression and syrinx size with outcome in patients with TCCS. | One year

CONTACTS AND LOCATIONS:
Overall Officials: Bizhan Aarabi, M.D., Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland Medical System, Baltimore, Maryland, United States